CLINICAL TRIAL: NCT06400251
Title: MATCH Treatment Subprotocol Z1K: Ipatasertib in Patients With Tumors With AKT Mutations
Brief Title: Testing Ipatasertib as Potentially Targeted Treatment in Cancers With AKT Genetic Changes (MATCH - Subprotocol Z1K)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2024-01194; NCI-2024-01194 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Z1K (Other: ECOG-ACRIN Cancer Research Group); EAY131-Z1K (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2024-05-03; First posted 2024-05-06 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Biopsy; Specimen Handling; ipatasertib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ipatasertib) (Experimental): Patients receive ipatasertib 400 mg PO QD on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo CT or MRI during screening and on study, as well as during follow-up as clinically necessary. Patients undergo biopsies and blood sample collection on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Ipatasertib; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Ipatasertib — Given PO
  Other Names: GDC 0068; GDC-0068; GDC0068; RG 7440; RG-7440; RG7440
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase II MATCH treatment trial tests how well ipatasertib works in treating patients with cancer that has certain genetic changes called AKT mutations. Ipatasertib is in a class of medications called protein kinase B (AKT) inhibitors. It may stop the growth of cancer cells and may kill them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE: Patients receive ipatasertib orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) during screening and on study, as well as during follow-up as clinically necessary. Patients undergo biopsies and blood sample collection on study.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol EAY131/ NCI-2015-00054 prior to registration to treatment subprotocol
* Patients must have an AKT mutation as determined via the MATCH Master Protocol
* Patients with breast cancer are excluded
* Patients with castration-resistant prostate cancer should maintain castrate levels of testosterone (i.e., with gonadotropin-releasing hormone (GnRH) agonists or through surgical castration). Patients are allowed to continue abiraterone acetate/prednisone with Ipatasertib if the patient just progressed on abiraterone acetate/prednisone
* Patients must not have known hypersensitivity to Ipatasertib or compounds of similar chemical or biologic composition
* Patients with known KRAS, NRAS, HRAS, or BRAF mutations are not eligible for this protocol, as these mutations may lead to limited response due to resistance
* Patients with diabetes or risk for hyperglycemia are eligible. Patients with diabetes mellitus should be on a stable dose of oral hypoglycemic agents for >= 4 weeks and appropriate diet. Patients with diabetes mellitus may enter the study unless any of the following exclusion criteria are fulfilled:

  * Baseline fasting glucose value of > 8.9 mmol/L or 160 mg/dL (fasting is defined as no calorific intake for at least 8 hours)
  * Patients not on a stable dose of oral hypoglycemic medication for >= 4 weeks and appropriate diet
  * Insulin required for routine diabetic management and control
  * More than two oral hypoglycemic medications required for routine diabetic management and control
  * Glycosylated hemoglobin (hemoglobin A1C) >= 7.5%
* Prior PI3K and mTOR inhibitors are allowed, including in the metastatic setting. Prior AKT inhibitors are excluded
* Patients with a history of inflammatory bowel diseases (Crohn's disease and ulcerative colitis) or active diverticulitis are not eligible
* Patients may not have received strong inhibitors or potent inducers or substrates of CYP3A4/5 within 2 weeks before the first dose of study treatment (3 weeks for St John's wort)
* In addition to the patient contraception requirements outlined in EAY131 MATCH Master Protocol, male patients must also refrain from donating sperm for the duration of study participation, and for 4 months after completion of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Kalinsky, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol Z1K was activated on July 25, 2019. Thirty-five patients were enrolled on EAY131-Z1K between August 8, 2019, and November 11, 2020. All patients were enrolled on the basis of the outside lab assay results.
Pre-assignment Details: Patients with tumors harboring E17K mutations in AKT1, 2, and 3, as well as Q79K and L52R mutations in AKT1, were eligible for sub-protocol Z1K. The mutation status was determined by an NCI-MATCH approved laboratory for all patients in this arm, they had to be confirmed by the NCI-MATCH central assay to be included in primary analysis.
Period: Overall Study
Arm/Group | Treatment (Ipatasertib)
Started | 35
Started Protocol Therapy | 34
Eligible and Treated | 32
Eligible, Treated and Mutation Status Confirmed (Primary efficacy analysis set) | 29
Completed | 0
Not Completed | 35
Not completed — Never Start Protocol Therapy | 1
Not completed — Ineligible | 2
Not completed — Mutation Status Not Confirmed | 3
Not completed — Disease Progression | 25
Not completed — Adverse Event | 1
Not completed — Complicating Disease | 1
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Patients who were eligible, started protocol therapy, and had mutation status confirmed at the analysis time were the analyzable patients
Arm/Group | Treatment (Ipatasertib)
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 63 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 22
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ipatasertib)
Number analyzed (Participants) | 29
percentage of participants | 24.1 [11.9 to 40.6]

2. Secondary Outcome: 6-month Progression Free Survival (PFS)
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ipatasertib)
Number analyzed (Participants) | 29
percentage of participants | 46.8 [30.9 to 61.2]

3. Secondary Outcome: Progression Free Survival
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Ipatasertib)
Number analyzed (Participants) | 29
months | 5.5 [3.6 to 12.9]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis. Thirty-four patients were included in the toxicity analysis (excluding one who did not receive treatment).
Arm/Group | Treatment (Ipatasertib)
All-Cause Mortality (participants affected / at risk) | 26/35
Serious Adverse Events (participants affected / at risk) | 13/34
Other Adverse Events (participants affected / at risk) | 27/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ipatasertib) (N=34)
Anemia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Fatigue (General disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Skin infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ipatasertib) (N=34)
Anemia (Blood and lymphatic system disorders) | 5
Fatigue (General disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 23
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 5
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 7
Creatinine increased (Investigations) | 6
Platelet count decreased (Investigations) | 2
Weight gain (Investigations) | 2
White blood cell decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT06400251/Prot_002.pdf
  • Informed Consent Form (2022-11-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT06400251/ICF_001.pdf